CLINICAL TRIAL: NCT00575757
Title: Relationship of Metabolic Abnormalities to Hepatic Steatosis in HIV
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: VCUHM10107; 1R03DK075416-01 (NIH)
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Steatohepatitis
Keywords: Steatosis; NASH
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sera, liver tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Primary: HIV infected with abnormal liver enzymes in the absence of HCV or HBV coinfections.

SUMMARY:
Because NASH is now recognized as a significant cause of cirrhosis with associated morbidity and mortality, its recognition as a long term complication of HAART is important to the management of those living with HIV.

DETAILED DESCRIPTION:
Abnormal liver enzymes are frequently seen in those with HIV. Although many of these individuals are co-infected with HBV or HCV, histology in HIV patients with abnormal liver enzymes in the absence of viral hepatitis has not been explored. HAART has significantly improved the survival in those living with HIV. However, components of HAART, particularly protease inhibitors (PIs) and certain nucleoside reverse transcriptase inhibitors (NRTIs), are frequently associated with metabolic abnormalities including insulin resistance (IR), dyslipidemias, fat redistribution and lipodystrophy (LD). Both IR and dyslipidemia are pathogenic mechanisms associated with nonalcoholic fatty liver disease (NAFLD) and non-alcoholic steatohepatitis (NASH) which often present as asymptomatic liver enzyme elevations. Because NASH is now recognized as a significant cause of cirrhosis with associated morbidity and mortality, its recognition as a long term complication of HAART is important to the management of those living with HIV. In our HIV population without HCV or HBV, there is a higher prevalence of abnormal liver enzymes (AST 21%, ALT 16%, ALP 43%) compared to the general population (ALT 8%) and is independently associated with PI use. The relationship of liver enzyme abnormalities to IR, dyslipidemias, and the development hepatic steatosis/NASH in HIV patients is unknown. We hypothesize that Liver enzyme abnormalities in HIV positive patients without viral hepatitis co-infections on HAART are due to hepatic steatosis related to PI use and that a subset of these individuals has NASH. The Specific Aims focus on HIV positive patients with abnormal liver enzymes in the absence of viral hepatitis co-infections, diabetes, or alcohol abuse to answer the following three questions: (1) What is the spectrum of NAFLD?; (2) How does the spectrum compare in those that are on a PI compare to those that are not; and (3) What are the independent predictive factors associated with hepatic steatosis and NASH? These studies will (1) provide novel data on the histology of HIV infected patients with abnormal liver enzymes in the absence of viral coinfections and their relationship to IR, LD, dyslipidemias, and HAART use and (2) provide the necessary pilot data for a multicenter R0-1 grant to study the long-term impact of HAART on the development of steatohepatitis and subsequent hepatic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* HIV antibody positive.
* Age > 18 years
* Abnormal liver chemistries (AST, ALT, and/or ALP) defined as between 1.25 -5 x ULN.

Exclusion Criteria:

* Hepatic decompensation: coagulopathy (prothrombin time prolonged > 2 seconds, INR > 1.5), ascites, hepatic encephalopathy, jaundice (serum conjugated bilirubin > 3.0)
* Thrombocytopenia (platelets < 80,000)
* Use of vitamin E, thiazolidinediones, metformin
* Use of medications associated with steatosis: amiodarone, methotrexate, corticosteroids, estrogen, and tamoxifen
* Renal failure (serum creatinine > 3.0)
* Diabetes mellitus
* Advanced HIV disease with life expectancy less than 1 year
* Alcohol use (> 40 grams/day in men and 20 grams/day in women)
* Presence of HCV RNA or HBV surface antigen
* Other liver diseases including alpha-1 antitrypsin (A1AT) deficiency, autoimmune hepatitis, hemochromatosis, Wilson's disease, HIV cholangiopathy, bacillary angiomatosis, lymphoma, and Kaposi's sarcoma
* Inability to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive with abnormal liver enzymes in the absence of HCV/HBV coinfections.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2007-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
What is the spectrum of NAFLD in HIV | 2 years

SECONDARY OUTCOMES:
How does the spectrum compare in those that are on a PI compare to those that are not. | 2 years
What are the independent predictive factors associated with hepatic steatosis and NASH? | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Sterling, MD MSc, Principal Investigator — VCU
Locations (1):
- Virgnia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Sterling RK, Smith PG, Brunt EM. Hepatic steatosis in human immunodeficiency virus: a prospective study in patients without viral hepatitis, diabetes, or alcohol abuse. J Clin Gastroenterol. 2013 Feb;47(2):182-7. doi: 10.1097/MCG.0b013e318264181d. PMID 23059409